CLINICAL TRIAL: NCT02939482
Title: A Prospective Study Comparison of Clinical Outcome After Different Rate Infusion in Caudal Epidural Steroid Injection
Brief Title: A Study Comparison of Clinical Outcome After Different Rate of Infusion in Caudal Epidural Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA 74/2559
Record Dates: First submitted 2016-10-15; First posted 2016-10-20 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Spinal Stenosis; Lumbosacral Spondylosis; Radiculopathy
MeSH Terms: conditions — Spinal Stenosis; Radiculopathy | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: 40 ml/min (Active Comparator): Triamcinolone acetonide (80 mg)/2 ml and normal saline solution 18 ml infusion in 0.5 min
  Interventions: Drug: Triamcinolone Acetonide and normal saline solution
- Group 2: 20 ml/min (Experimental): Triamcinolone acetonide (80 mg)/2 ml and normal saline solution 18 ml infusion in 1 min
  Interventions: Drug: Triamcinolone Acetonide and normal saline solution

INTERVENTIONS:
Drug: Triamcinolone Acetonide and normal saline solution — 80 mg/2 ml Triamcinolone Acetonide and 18 ml normal saline solution

SUMMARY:
The purpose of this study is to determine the effects of different rates of Caudal Epidural Steroid Injection (CESI) on clinical outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

* lumbosacral spinal stenosis with radiculopathy
* no improvement after conservative treatment for 6 weeks

Exclusion Criteria:

* previous CESI or spinal surgery
* skin infection at injection site
* uncontrolled diabetes mellitus
* abnormal coagulogram
* vertebral fracture
* previous history of allergy to steroid or anesthetic agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Visual Analogue Scale at 2, 6, 12 weeks | 2, 6, 12 weeks
Change from baseline Roland 5-point pain scale at 2, 6, 12 weeks | 2, 6, 12 weeks
Change from baseline Standing tolerance test at 2, 6, 12 weeks | 2, 6, 12 weeks
Change from baseline Walking tolerance test at 2, 6, 12 weeks | 2, 6, 12 weeks
Change from baseline Patient satisfaction scale at 2, 6, 12 weeks | 2, 6, 12 weeks

SECONDARY OUTCOMES:
Complication of Caudal Epidural Steroid Injection | 2, 6, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Watts RW, Silagy CA. A meta-analysis on the efficacy of epidural corticosteroids in the treatment of sciatica. Anaesth Intensive Care. 1995 Oct;23(5):564-9. doi: 10.1177/0310057X9502300506. PMID 8787255
- [Result] Botwin KP, Gruber RD, Bouchlas CG, Torres-Ramos FM, Sanelli JT, Freeman ED, Slaten WK, Rao S. Fluoroscopically guided lumbar transformational epidural steroid injections in degenerative lumbar stenosis: an outcome study. Am J Phys Med Rehabil. 2002 Dec;81(12):898-905. doi: 10.1097/00002060-200212000-00003. PMID 12447088
- [Result] Kraiwattanapong C, Wechmongkolgorn S, Chatriyanuyok B, Woratanarat P, Udomsubpayakul U, Chanplakorn P, Keorochana G, Wajanavisit W. Outcomes of fluoroscopically guided lumbar transforaminal epidural steroid injections in degenerative lumbar spondylolisthesis patients. Asian Spine J. 2014 Apr;8(2):119-28. doi: 10.4184/asj.2014.8.2.119. Epub 2014 Apr 8. PMID 24761192